CLINICAL TRIAL: NCT04133636
Title: A Phase 2, Multicohort Open-Label Study of JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against BCMA in Subjects With Multiple Myeloma
Brief Title: A Study of JNJ-68284528, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against B-cell Maturation Antigen (BCMA) in Participants With Multiple Myeloma
Acronym: CARTITUDE-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108581; 68284528MMY2003 (Other: Janssen Research & Development, LLC); 2018-004124-10 (EudraCT Number); 2023-506587-13-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Cellular Therapy; CAR-T Therapy; BCMA CAR-T
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; daratumumab; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-68284528 (Experimental): Single group assignment-Post lymphodepletion, JNJ-68284528 single infusion given to Part A participants: Cohort A(Progressive disease post 1-3 prior lines of therapy), Cohort B(Early relapse post front-line), Cohort C(Relapsed/refractory multiple myeloma post PI, IMiD,anti-CD38,anti-BCMA therapy), Cohort D(Less than CR post ASCT front-line therapy, some participants will receive JNJ-68284528 then lenalidomide), Cohort F(Newly diagnosed multiple myeloma [NDMM], standard risk [International Staging System Stage I/II] and post initial therapy); Cohort E(NDMM,transplant not planned,high risk disease) will first receive quadruplet induction regimen of daratumumab,bortezomib,lenalidomide and dexamethasone(D-VRd) then lymphodepletion and JNJ-68284528 then consolidation regimen of lenalidomide. Part B:Cohort G(NDMM,transplant not planned) will receive daratumumab, lenalidomide and dexamethasone followed by cilta-cel; Cohort H(NDMM,transplant-eligible) will receive D-VRd followed by cilta-cel.
  Interventions: Drug: JNJ-68284528; Drug: Lenalidomide; Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: JNJ-68284528 — Participants in Cohorts A,B,C, D, E, F, G, and H will receive JNJ-68284528 intravenously.
  Other Names: Ciltacabtagene autoleucel (cilta-cel)
Drug: Lenalidomide — Some participants in Cohort D and all participants in Cohorts E, G, and H will also receive lenalidomide capsules orally.
Drug: Daratumumab — Participants in Cohorts E, G, and H will also receive daratumumab subcutaneous (SC) injection.
Drug: Bortezomib — Participants in Cohorts E and H will also receive bortezomib subcutaneously.
Drug: Dexamethasone — Participants in Cohorts E, G, and H will also receive dexamethasone orally or intravenously.

SUMMARY:
The purpose of this study is to evaluate the overall minimal residual disease (MRD) negative rate of participants who receive JNJ-68284528.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Received a minimum of 1 to a maximum of 3 prior lines of therapy including a proteasome inhibitor (PI) and immunomodulatory therapy (IMiD), and lenalidomide refractory per International Myeloma Working Group (IMWG) guidelines
* Cohort B: Received one line of prior therapy including a PI and an IMiD, and disease progression per IMWG criteria less than or equal to (<=) 12 months after treatment with autologous stem cell transplantation (ASCT) or <=12 months from the start of anti-myeloma therapy for participants who have not had an ASCT
* Cohort C: Previously treated with a PI, an IMiD, an anti-CD38 monoclonal antibody and B-cell maturation antigen (BCMA)-directed therapy
* Cohort D: Newly diagnosed multiple myeloma per IMWG with a history of 4 to 8 total cycles of initial therapy, including induction, high-dose therapy, and ASCT with or without consolidation
* Cohort E: Have newly diagnosed multiple myeloma without prior therapy (one cycle of prior therapy before enrollment is acceptable) and classified as high risk defined as either: 1) International Staging System (ISS) stage III criteria, Beta 2 microglobulin greater than or equal to (>=) 5.5 milligrams per liter (mg/L) (via local or central laboratory assessment) or 2) high risk cytogenetic features del(17/17p), t (14;16), t(14;20), 1q amplification (at least 4 total copies) in at least 20 percent (%) of the total plasma cell population
* Cohort F:
* Participant must have a documented efficacy response of very good partial response (VGPR) or better, without progressive disease prior to enrollment, as assessed per IMWG 2016 criteria
* Received initial therapy as specified below. The dose/schedule of cycles administered will be as per standard of care. It is acceptable for up to 1 cycle of the protocol-specified regimens to be missing one of the listed agents (example, held due to toxicity). Acceptable combinations include: At least 5 to 8 cycles of initial therapy with daratumumab, bortezomib, lenalidomide and dexamethasone (D-VRd). The dose/schedule of cycles administered will be as per standard of care or; at least 4 to 8 cycles of initial therapy with daratumumab, lenalidomide and dexamethasone (D-Rd) or; at least 4 to 8 cycles of initial therapy with a carfilzomib-based triplet or quadruplet regimen
* Cohort G: Not considered for high-dose chemotherapy with autologous stem cell transplantation (ASCT) due to: a) Ineligibility due to advanced age; or b) Ineligibility due to presence of comorbid condition(s) likely to have a negative impact on tolerability of high-dose chemotherapy with ASCT; or c) Subject refusal of high-dose chemotherapy with ASCT as initial treatment
* Cohort H: Considered a candidate for high-dose chemotherapy with ASCT as initial treatment
* Cohorts A, B, C, E, G, H:
* Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 1.0 gram per deciliter (g/dL) or urine M-protein level >=200 milligrams (mg)/24 hours
* Light chain multiple myeloma in whom only measurable disease is by serum free light chain (FLC) levels in the serum: Serum immunoglobulin FLC >=10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio
* Cohort A: For participants with neither serum nor urine measurable disease, baseline positron emission tomography/ computed tomography (PET/CT) or whole -body magnetic resonance imaging (MRI) may be used to satisfy the measurable disease criteria. A minimum of one lesion with a bi-dimensional measurement of at least 1 centimeter (cm)*1 cm is required
* Cohorts B, C: For participants with neither serum nor urine measurable disease, baseline positron emission tomography/ computed tomography (PET/CT) or whole body magnetic resonance imaging (MRI) may be used to satisfy the measurable disease criteria
* Cohorts A, B, C, D, E, F, G, H: Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1

Exclusion Criteria:

* Cohorts A, B, D, F: Any therapy that is targeted to BCMA
* Cohorts A, B, C, D, F: Prior treatment with chimeric antigen receptor T (CAR-T) therapy directed at any target
* Cohorts A, B, C, D, F:
* Ongoing toxicity from previous anticancer therapy must resolve to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Received a cumulative dose of corticosteroids equivalent to >=70 mg of prednisone within the 7 days (Cohort A, B, C, F) or 14 days (Cohort D) prior to apheresis
* Serious underlying medical condition, such as (a) evidence of active viral or bacterial infection requiring systemic antimicrobial therapy, or uncontrolled systemic fungal infection; (b) active autoimmune disease or a history of autoimmune disease within 3 years; (c) overt clinical evidence of dementia or altered mental status; (d) any history of Parkinson's disease or other neurodegenerative disorder
* Cohorts A, B, C, D, E, F: Known active, or prior history of central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of multiple myeloma
* Cohorts F, G, and H: Active malignancies (that is, progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are: a) non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured; b) skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured; c) non-invasive cervical cancer treated within the last 24 months that is considered completely cured; d) localized prostate cancer (N0M0): with a Gleason score of greater than or equal to (=>)6, treated within the last 24 months or untreated and under surveillance, with a Gleason score of 3+4 that has been treated more than 6 months prior to full study screening and considered to have a very low risk of recurrence, or history of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence, e) breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence; f) malignancy that is considered cured with minimal risk of recurrence
* Cohorts E, G, and H: Frailty index of >= 2 according to Myeloma Geriatric Assessment score

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2029-09-03 (Estimated)

PRIMARY OUTCOMES:
Cohorts A, B, C, D, E, and F: Percentage of Participants with Negative Minimal Residual Disease (MRD) | At least 1 year after JNJ-68284528 infusion on Day 1
  MRD negative rate is the percentage of participants who achieve MRD negative status by evaluation of bone marrow aspirate as defined by the International Myeloma Working Group (IMWG) criteria.
Cohorts G and H: Percentage of Participants with Sustained MRD Negative Complete Response (CR) | At least 1 year after JNJ-68284528 infusion on Day 1
  Sustained MRD-negative CR is defined as participants with CR or better who sustain MRD-negative status, as determined by next-generation sequencing (NGS) or next generation flowcytometry (NGF) with sensitivity of 10^-5, for at least 12 months without any examination showing MRD positive status or progressive disease in between.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years and 6 months
  ORR is defined as the percentage of participants who achieve a partial response (PR) or better according to the IMWG criteria.
Cohorts A, B, C, D, E, and F: VGPR or Better Rate | Up to 2 years and 6 months
  The VGPR or better rate (stringent complete responses [sCR] + complete response [CR] + VGPR), defined as the percentage of participants achieving VGPR or better response according to IMWG criteria during or after the study treatment.
Cohorts A, B, C, D, E, and F: Clinical Benefit Rate (CBR) | Up to 2 years and 6 months
  CBR is defined as the percentage of participants who achieve ORR (sCR + CR + VGPR + PR) + minimal response (MR) according to the IMWG criteria.
Duration of Response (DOR) | Up to 2 years and 6 months
  DOR will be calculated among responders from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG criteria.
Time to Response (TTR) | Up to 2 years and 6 months
  TTR is defined as the time from the date of the initial infusion of JNJ-68284528 and the first efficacy evaluation that the participant has met all criteria for PR or better.
Cohorts A, B, C, D, E, and F: MRD Negative Rate at 12 Months for Participants who Achieve a Complete Response (CR) | 12 months
  MRD negative rate at 12 months for participants who achieved a complete response (CR) is defined as the percentage of participants who are MRD negative by bone marrow aspirate and meet the IMWG criteria for CR at 12 months after initial dose of JNJ-68284528 and before disease progression or starting subsequent therapy including retreatment of JNJ-68284528.
Time to MRD Negativity | Up to 2 years and 6 months
  Time to MRD negativity will be calculated in participants who are MRD negative by bone marrow aspirate from the date of the initial infusion of JNJ-68284528 to the initial date of reaching the MRD negative status.
Duration of MRD Negativity | Up to 2 years and 6 months
  Duration of MRD negativity will be calculated among participants who are MRD negative by bone marrow aspirate from the date of initial MRD negativity to the date when MRD is detected at the same threshold (10^-5).
Cohorts A, B, C, D, E, and F: MRD Negative Rate Across Clinical Response | Up to 2 years and 6 months
  MRD negative rate across clinical response groups will be assessed for all participants who achieved a complete response (CR) or stringent complete response (sCR) or very good partial response (VGPR) according to the IMWG criteria during or after the study treatment. MRD negative rate is defined as the percentage of participants who have negative MRD by bone marrow aspirate at any timepoint.
Number of Participants with Adverse Events by Severity | Up to 2 years and 6 months
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), with the exception of cytokine release syndrome (CRS), and immune effector cell-associated neurotoxicity syndrome (ICANS). CRS and ICANS will be evaluated according to the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading.
Number of Participants with Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 2 years and 6 months
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Laboratory Abnormalities | Up to 2 years and 6 months
  Number of participants with laboratory abnormalities will be reported.
Number of Participants with Vital Signs Abnormalities | Up to 2 years and 6 months
  Number of participants with vital signs abnormalities will be reported.
Cohorts A, B, C, D, E, and F: Levels of B-Cell Maturation Antigen (BCMA) Expressing Cells and Soluble BCMA | Up to 1 year
  Levels of expression of BCMA-expressing plasma cells in the bone marrow as well as the level of soluble BCMA in blood will be reported.
Cohorts A, B, C, D, E, and F: Systemic Inflammatory Cytokine Concentrations | Up to 1 year
  Blood cytokine concentrations (Interleukin [IL]-6, IL-15, IL-10, and Interferon [IFN-gamma]) will be measured for biomarker assessment.
Cohorts A, B, C, D, E, and F: Levels of JNJ-68284528 T Cell Expansion (proliferation), and Persistence | Up to 1 year
  Levels of JNJ-68284528 T cell expansion (proliferation), and persistence via monitoring CAR-T positive cell counts and CAR transgene level will be reported.
Cohorts A, B, C, D, E, and F: Number of Participants with Anti-JNJ-68284528 Antibodies | Up to 1 year
  Number of participants exhibiting anti-drug antibodies for JNJ-68284528 will be reported.
Cohorts G and H: Percentage of Participants with Complete Response (CR) or Better | Up to 2 years 6 months
  CR or better is defined as the percentage of participants achieving CR or sCR prior to subsequent antimyeloma therapy in accordance with the IMWG criteria during or after the study treatment.
Cohorts G and H: Percentage of Participants with MRD-negative CR or sCR | Up to 2 years 6 months
  MRD-negative CR/sCR is defined as the percentage of participants who achieve MRD-negative status, as determined by NGS/NGF with sensitivity of 10^-5, at any time after enrollment and prior to progressive disease or subsequent antimyeloma therapy and who achieve CR/sCR or better.
Cohorts G and H: Progression-free Survival on Next-line Therapy (PFS2) | Up to 2 years and 6 months
  PFS2 is defined as the time interval between the start of study treatment and date of event, which is defined as death from any cause or PD as assessed by investigator that starts after the next line of therapy, whichever occurs first.
Cohorts G and H: Overall Survival (OS) | Up to 2 years and 6 months
  OS is defined as the time from the start of study treatment to the date of the participant's death.
Cohorts G and H: Progression-free Survival (PFS) | Up to 2 years and 6 months
  PFS is defined as the time from the start of study treatment to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Cohorts G and H: Number of Participants with Measurable Replication Competent Lentivirus (RCL) in Whole Blood | Up to 2 years and 6 months
  Number of participants with measurable RCL in whole blood will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (33):
  - University Of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- France (3):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - C.H.U. Hotel Dieu - France, Nantes
  - Hopital Saint Louis, Paris
- Germany (2):
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitatsklinikum Wurzburg, Würzburg
- Israel (2):
  - Sheba Medical Center Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Spain (2):
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Cohen AD, Mateos MV, Cohen YC, Rodriguez-Otero P, Paiva B, van de Donk NWCJ, Martin T, Suvannasankha A, De Braganca KC, Corsale C, Schecter JM, Varsos H, Deraedt W, Wang L, Vogel M, Roccia T, Xu X, Mistry P, Zudaire E, Akram M, Nesheiwat T, Pacaud L, Avivi I, San-Miguel J. Efficacy and safety of cilta-cel in patients with progressive multiple myeloma after exposure to other BCMA-targeting agents. Blood. 2023 Jan 19;141(3):219-230. doi: 10.1182/blood.2022015526. PMID 36095849
- See also: Related Info — https://myeloma.sparkcures.com/trial/1039/nct04133636?utm_source=bhm&utm_medium=digital&utm_campaign=cartitude2